CLINICAL TRIAL: NCT02761889
Title: Hypofractionated Image-Guided Radiotherapy (IGRT) With Organ Motion Mitigation and Urethral Sparing for Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Principal Investigator, Carlo Greco, MD, Director of Clinical Research, Fundacao Champalimaud
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYPO
Record Dates: First submitted 2016-04-26; First posted 2016-05-04 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Adenocarcinoma of the Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IGRT 45 Gy in 5 fractions of 9 Gy (Experimental): Patients will be treated using volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. Patients will be treated with 45 Gy in five fractions of 9 Gy over 5 consecutive days.
  Interventions: Radiation: IGRT 45 Gy in 5 fractions of 9 Gy; Procedure: Image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT); Device: Rectal balloon with air filling; Device: Urethral catheter loaded with beacon transponders

INTERVENTIONS:
Radiation: IGRT 45 Gy in 5 fractions of 9 Gy — Previously untreated patients with prostate cancer will be treated with 45 Gy in five fractions of 9 Gy over 5 consecutive days.
Procedure: Image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) — Patients enrolled in the study will undergo IGRT-VMAT with state-of-the-art treatment-planning and quality assurance procedures with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility.
Device: Rectal balloon with air filling — A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility.
Device: Urethral catheter loaded with beacon transponders — A urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking.

SUMMARY:
The present study evaluates the clinical outcomes following definitive ultra-high dose per fraction external beam radiation therapy delivered in patients with organ-confined adenocarcinoma of the prostate.

Patients enrolled in the study will undergo image-guided, volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) with state-of-the-art treatment-planning and quality assurance procedures with emphasis on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility, while a urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking. Previously untreated patients with prostate cancer will be treated with 45 Gy in five fractions of 9 Gy over 5 consecutive days.

Patients will be followed at one month post-treatment and every 3 months for up to 12 months (+/- 4 weeks) and every 6 months (+/- 6 weeks) thereafter. Acute and late toxicity evaluations will focus, though not exclusively, on urinary, rectal and sexual functions and will be assessed through validated Expanded Prostate Cancer Index Composite (EPIC), International prostate symptom score (IPSS) and International index of erectile function (IIEF) questionnaires. Serum Prostate Specific Antigen (PSA) values will be drawn on the same schedule as clinical follow-up. Patients will be continuously monitored for a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed study specific informed consent form;
* Histologic confirmation of adenocarcinoma of the prostate by biopsy;
* Previous hormonal therapy is allowed (but not required);
* No direct evidence of regional or distant metastases after appropriate staging studies;
* Age ≥ 40;
* Performance Status 0-2;
* American Urological Association (AUA) score must be ≤ 20 (alpha blockers allowed);
* Computerized Tomography (CT) or Ultrasound-based volume estimation of prostate gland ≤ 150 grams.

Exclusion Criteria:

* Metastatic disease from prostate cancer on imaging studies MRI evidence of radiographic T3, T4;
* Previous pelvic radiotherapy;
* Previous surgery for prostate cancer;
* Previous hormonal therapy given for more than 6 months prior to therapy;
* History of Crohn's Disease or Ulcerative Colitis;
* Previous significant obstructive symptoms;
* Significant psychiatric illness;
* Severe, active co-morbidity as defined in section 3.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-related grade 3 gastrointestinal or genitourinary toxicity adverse events as assessed by NCI v3.0. | 5 years
Changes in PSA biochemical parameter measurements (Phoenix Definition). | 5 years
Expanded Prostate Cancer Index Composite (EPIC) Questionnaire to measure quality of life. | 5 years
International Index of Erectile Function (IIEF) Questionnaire to measure quality of life. | 5 years
International Prostate Symptom Score (IPSS) Questionnaire to measure quality of life. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Greco, MD, Principal Investigator — Fundacao Champalimaud
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greco C, Pares O, Pimentel N, Louro V, Nunes B, Kociolek J, Marques J, Fuks Z. Early PSA density kinetics predicts biochemical and local failure following extreme hypofractionated radiotherapy in intermediate-risk prostate cancer. Radiother Oncol. 2022 Apr;169:35-42. doi: 10.1016/j.radonc.2022.02.016. Epub 2022 Feb 18. PMID 35189157